CLINICAL TRIAL: NCT05264246
Title: Evaluation of an Anti-Shivering Protocol for Targeted Temperature Management Following Cardiac Arrest
Brief Title: Evaluation of an Anti-Shivering Protocol Cardiac Arrest
Status: Terminated | Type: Observational
Why Stopped: PI requested to close the study. No study activity since 2021 and no intent to publish results.
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 042.PHA.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This will be a single center, retrospective, before-and-after, chart review of all patients undergoing TTM between June 1, 2017 and May 31, 2021 at MDMC. Initiation of the new TTM protocol occurred on April 22, 2019.

DETAILED DESCRIPTION:
This will be a single center, retrospective, before-and-after, chart review of all patients undergoing TTM between June 1, 2017 and May 31, 2021 at MDMC. Initiation of the new TTM protocol occurred on April 22, 2019. To allow for an adequate washout period, patients who were initiated on TTM before April 22, 2019 will be in the "before" group and patients initiated on TTM on or after June 1, 2019 will be in the "after" group. Patients will be identified based on electronic medical records search of order sets utilized in TTM and confirmed with manual chart review. Statistical analysis will be performed as detailed below.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of cardiac arrest
* Initiation of TTM via Arctic Sun® device

Exclusion Criteria:

* Initiation of TTM > 12 hours after cardiac arrest
* Receiving NMBs for an indication other than TTM
* Early termination of TTM (less than 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to conduct the retrospective chart review of all patients identified during the study period (from June 1, 2017 to May 31, 2021) that meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
NMB usage | June 1, 2017 - May 31, 2021
  vecuronium or cisatracurium

SECONDARY OUTCOMES:
NMB usage | June 1, 2017 - May 31, 2021
  Proportion of patients that required any vecuronium boluses
  Number of vecuronium boluses administered
  Proportion of patients that required initiation of cisatracurium infusion
Patients discharged home | June 1, 2017 - May 31, 2021
  Proportion of patients discharged home
Patients with a breakthrough fever (temperature > 38°C) in the first 72 hours of TTM initiation | First 72 hours of TTM initiation
  Proportion of patients with a breakthrough fever (temperature > 38°C) in the first 72 hours of TTM initiation
Proportion of patients cooled to 33°C versus 36°C | June 1, 2017 - May 31, 2021
  number of patients at desired temperature range
Time to target temperature from initiation of TTM | June 1, 2017 - May 31, 2021
  time in minutes
ICU length of stay | June 1, 2017 - May 31, 2021
  number of days

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Reiter, PharmD, Principal Investigator — Methodist
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States